CLINICAL TRIAL: NCT02583997
Title: Non-closure of Alveoli After Avulsion of Wisdom Teeth: a Randomized, Open, Multicenter Trial
Brief Title: Non-closure of Alveoli After Avulsion of Wisdom Teeth
Acronym: AlvéCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2014/PL-01; 2014-A00512-45 (Other: ANSM)
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2018-08

CONDITIONS: Wisdom Tooth Avulsion
Keywords: To suture or not to suture....; Tooth extraction; Third molar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine third molar extraction (Active Comparator): Patients randomized to this arm will have all four wisdom teeth removed according to usual, standard care (i.e. with suturing of the lower alveoli).
  Intervention: Suturing of lower alveoli
  Interventions: Procedure: Suturing of lower alveoli
- Third molar extraction without suturing (Experimental): Patients randomized to this arm will have all four wisdom teeth removed according to usual, standard care, except that the resulting alveoli will not be sutured.
  Intervention: Non suturing of lower alveoli
  Interventions: Procedure: Non suturing of lower alveoli

INTERVENTIONS:
Procedure: Suturing of lower alveoli — After extraction of wisdom teeth, the lower alveoli are sutured closed.
  Arms: Routine third molar extraction
Procedure: Non suturing of lower alveoli — After extraction of wisdom teeth, no alveoli are sutured closed.
  Arms: Third molar extraction without suturing

SUMMARY:
The main objective of this study is to evaluate postoperative pain (measured by visual analogue scale (VAS) on day 2 post surgery) in patients operated for avulsion of four wisdom teeth under general anesthesia and for whom the resulting alveoli were NOT sutured versus a similar group of patients undergoing standard care (suturing for lower alveoli).

DETAILED DESCRIPTION:
The secondary objectives of this study are to compare the following between the two study arms:

A. Pain at day 31 B. Operative time C. Edema D. Trismus E. The occurrence of complications F. Alveolar flap healing G. The impact of smoking on the occurrence of complications H. The consumption of analgesics and use of local pain remedies I. Impact on quality of life

ELIGIBILITY:
Inclusion Criteria:

* The patient was correctly informed about the implementation of the study, its objectives, constraints and patient rights
* The patient gave his/her free and informed signed consent
* For patients under 18 years of age, the patient's parents (or legal guardian) must have given their free and informed signed consent
* The patient must be affiliated with or the recipient of a health insurance program
* The patient is available for 31 days of follow-up
* The patient is a candidate for avulsion of all 4 wisdom teeth under general anesthesia

Exclusion Criteria:

* The patient is participating in another study
* The patient has participated in another study in the last 3 months
* The patient is in an exclusion period is determined by a previous study
* The patient is an adult under guardianship
* The patient is under judicial protection
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* For patients under 18 years of age, his/her parents (or legal guardian) refuse to sign the consent
* The patient is pregnant, breastfeeding or parturient
* The patient has a contra-indication (or an incompatible combination therapy) for a treatment in this study
* The patient is taking antiplatelet agents
* The patient is taking anticoagulants
* The patient has a coagulation disorder
* The patient suffers from immunosuppression
* The patient's wisdom teeth are in a normal, functional, healthy position
* Other orofacial surgical procedures are planned during the study period
* Active pericoronitis

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Visual analog scale for pain. | Day 2
  Surgery is on day 0.

SECONDARY OUTCOMES:
Visual analog scale for pain. | Day 0
Visual analog scale for pain. | Day 31
Operative time | Day 0
  From time of first incision to moment when sterile fields are removed.
Edema | Day 0: post-op.
  ((D-Dbaseline)/Dbaseline)*100
  Where D =[(the distance from the lobe of the left ear to the left labial commissure)+(the distance from the lobe of the right ear to the right labial commissure)]/2. D is measured in mm. D evaluates edema.
  The Dbaseline measure is made just before surgery.
Edema | Day 2
  ((D-Dbaseline)/Dbaseline)*100
  Where D =[(the distance from the lobe of the left ear to the left labial commissure)+(the distance from the lobe of the right ear to the right labial commissure)]/2. D is measured in mm. D evaluates edema.
  The Dbaseline measure is made just before surgery.
Edema | Day 31
  ((D-Dbaseline)/Dbaseline)*100
  Where D =[(the distance from the lobe of the left ear to the left labial commissure)+(the distance from the lobe of the right ear to the right labial commissure)]/2. D is measured in mm. D evaluates edema.
  The Dbaseline measure is made just before surgery.
Trismus | Day 0: post-op.
  ((T-Tbaseline)/Tbaseline)*100
  Where T = A measure of maximum mouth opening in mm ; T evaluates trismus.
  The Tbaseline measure is made just before surgery.
Trismus | Day 2
  ((T-Tbaseline)/Tbaseline)*100
  Where T = A measure of maximum mouth opening in mm ; T evaluates trismus.
  The Tbaseline measure is made just before surgery.
Trismus | Day 31
  ((T-Tbaseline)/Tbaseline)*100
  Where T = A measure of maximum mouth opening in mm ; T evaluates trismus.
  The Tbaseline measure is made just before surgery.
The occurrence of complications | Day 0
  The occurrence of at least one complication among the following with at least one of the 4 teeth:
  * Hemorrhage: occurrence of continuous or intermittent bleeding from the socket immediately after extraction of the wisdom tooth or later on
  * Infection: occurrence of purulent discharge, a collection of pus or cellulitis at the surgical site
  * Dry alveolitis: presence of an empty socket with a whitish, atonal bone, giving off a foul odor and very sensitive
  * Suppurative alveolitis: presence of granulomatous tissue, bleeding and pus in the socket. The latter are accompanied by pain, trismus, low-grade fever, and regional lymphadenopathy.
For the experimental arm: good flap healing? (ie no attachment loss at the second molar) (per tooth). | Day 0
For the experimental arm: good flap healing? (ie no attachment loss at the second molar) (per tooth). | Day 2
For the experimental arm: good flap healing? (ie no attachment loss at the second molar) (per tooth). | Day 31
The consumption of analgesics | Day 0
The consumption of analgesics | Day 2
The consumption of analgesics | Day 31
The General Oral Health Assessment Index questionnaire | Day 0
The General Oral Health Assessment Index questionnaire | Day 31

OTHER OUTCOMES:
Age | Baseline (day 0)
Gender | Baseline (day 0)
Body mass index | Baseline (day 0)
Number of cigarettes smoked per day | Day 0
Number of cigarettes smoked per day | Day 2
Number of cigarettes smoked per day | Day 31
Proximity of the M3 nerve for each tooth | Baseline (day 0)
Winter classification for each tooth | Baseline (day 0)
Delay between surgery and the first post-operative measure (e.g. for edema or trismus) | Day 0
Surgical indication (i.e. why the avulsion is being performed). | Baseline (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lapeyrie, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - CHRU de Montpellier - Hôpital Gui de Chauliac, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - CH de Perpignan - Hôpital Saint Jean, Perpignan

REFERENCES:
- [Result] Takadoum S, Douilly G, de Boutray M, Kabani S, Maladiere E, Demattei C, Lapeyrie P. Sutureless socket technique after removal of third molars: a multicentric, open, randomized controlled trial. BMC Oral Health. 2022 Jun 26;22(1):256. doi: 10.1186/s12903-022-02287-y. PMID 35754043